CLINICAL TRIAL: NCT06817070
Title: Dietary Patterns, Physical Activity, and Nutritional Challenges Among Mexican Adults During the COVID-19 Pandemic: A Cross-Sectional Study
Brief Title: Diet, Exercise, and Nutrition Challenges in Mexican Adults During COVID-19: A Study
Acronym: UDEM Covid19
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Queretaro (Other)
Collaborators: Universidad de Monterrey (Other); Tecnologico de Monterrey (Other); Universidad de Granada (Other)
Responsible Party: Principal Investigator, Ivan Luzardo-Ocampo, Professor-Researcher, Universidad Autonoma de Queretaro
Other Study IDs: UDEM-AGOC21
Record Dates: First submitted 2025-02-06; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: COVID19 Disease
Keywords: SARS Cov-2; Frequency of intake; dietary patterns; ultraprocessed foods; mexican population

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- General Study Group: Overall participants having either underweight, normal weight, overweight, or the 3 obesity types
  Interventions: Diagnostic Test: Food Consumption survey

INTERVENTIONS:
Diagnostic Test: Food Consumption survey — A comprehensive survey was created using Google Forms® to collect sociodemographic, clinical, anthropometric, dietary data, and physical activity information from participants across most Mexican states. All self-administered surveys began with informed consent and were distributed via instant messaging (WhatsApp), social networks (Facebook, Twitter), and email using a snowball sampling method. Sociodemographic data included age, gender, and residence, while anthropometric data covered weight, height, and physical activity. Food intake was assessed using a 48-item semi-quantitative tool based on the National Health and Nutrition Survey 2021, with participants reporting the frequency and quantity of food consumed on a Likert scale. Responses were converted to daily consumption values and caloric intake using the Mexican System of Foods and Equivalents. Foods and beverages were categorized into twelve groups: six healthy (fruits, vegetables, legumes, natural dairy, white meat, nuts, and
  Other Names: Anthropometric characteristics

SUMMARY:
The COVID-19 pandemic was particularly devastating in developing countries such as Mexico, where the nation reported some of the highest COVID-19 cases and a high prevalence of obesity. This study aimed to evaluate the food consumption among Mexican adults during the COVID-19 pandemic. A cross-sectional study was conducted, involving 1,082 Mexican adults recruited through online invitations containing a link to complete a survey. A 48-item questionnaire was designed to assess the frequency of food consumption and sociodemographic characteristics in a semi-quantitative manner. A retrospective instrument was used to evaluate physical activity (days/week and duration).

DETAILED DESCRIPTION:
The COVID-19 pandemic had a particularly harsh impact on developing countries like Mexico, which reported some of the highest numbers of COVID-19 cases and a significant prevalence of obesity. This study aimed to examine the eating habits of Mexican adults during the COVID-19 pandemic. A cross-sectional survey was conducted, involving 1,082 Mexican adults who were recruited via online invitations that included a link to complete a questionnaire. A 48-item survey was created to evaluate the frequency of food consumption and sociodemographic factors semi-quantitatively. Physical activity was assessed using a retrospective tool to measure the frequency and duration of exercise per week.

The main discovery identified two dietary patterns: industrialized and healthy. The industrialized dietary pattern was more common and included the consumption of sugary dairy products, sugary drinks, alcoholic beverages, sweets, fried foods, and both red and processed meats. Men consumed significantly more ultra-processed foods (22.5%) compared to women (15.45%) based on a 2000 kcal diet. In addition, participants did not meet the recommended intake levels for fruits, vegetables, legumes, and natural dairy products. Intake of sugary drinks was three times higher than recommended for both genders. Regarding physical activity, only 29.7% of participants reported engaging in adequate physical activity.

The study also highlighted insufficient consumption of nuts and an excessive intake of red and processed meats. It underscored the necessity for intervention and educational initiatives to improve dietary choices, particularly among younger populations.

ELIGIBILITY:
Inclusion Criteria: Additional to the age, people living in Mexico during the COVID pandemics.

Exclusion Criteria: People who did not live in Mexico during the COVID pandemics

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People living in Mexico during the pandemic, from all the states and genders.
Sampling Method: Non-Probability Sample
Enrollment: 1082 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Sociodemographics | 2 months
  The survey yielded a sample of 1,082 participants. Women made up 66% of the respondents. The majority of participants were in the 18 to 24-year-old age group (48.9%), followed by those aged 25 to 34 (15.8%). As for BMI, 64% of participants reported having a normal BMI. Additionally, 47.9% indicated they led a sedentary lifestyle, whereas only 29.7% reported engaging in optimal physical activity.
Dietary Patterns | 2 months
  Two dietary patterns were identified in the study. The first, termed the "industrialized diet," is characterized by high consumption of natural dairy products, white meats, processed dairy products with added sugar, red and processed meats, alcoholic beverages, sugary drinks, confectionery, sweets, snacks, and fried foods. The second, known as the "healthy dietary pattern," includes high consumption of fruits, vegetables, legumes, natural dairy products, white meats, and nuts. These patterns explained 43.33% of the total variance in the participants' diets.

CONTACTS AND LOCATIONS:
Overall Officials: Anayansi Escalante-Aburto, Ph. D., Study Chair — Tecnologico de Monterrey
Locations (1):
- Universidad de Monterrey, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a research manuscript.
Supporting Information: Study Protocol
Time Frame: June 2025 to June 2027
Access Criteria: Researchers and academics
URL: https://scholar.google.es/citations?user=r3VZ8HcAAAAJ&hl=es&oi=ao